CLINICAL TRIAL: NCT04396080
Title: Prospective Clinical Trial of Onlay-carrying Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H1543943843337
Record Dates: First submitted 2020-05-11; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-03

CONDITIONS: Success; Survival Rate; Clinical Performance

STUDY DESIGN:
Intervention Model Description: Patients who require it, will be treated with posterior partial restorations. That will be the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Onlays behaviour depending on materials (Experimental): Patients who require it as treatment option will be treated with posterior partial restorations, and will have clinical follow-up to obtain a comparison of the behavior of subsequent restorations based on the material.
  Interventions: Procedure: Partial restoration in posterior teeth

INTERVENTIONS:
Procedure: Partial restoration in posterior teeth — Teeth in need of onlays that will be treated with this type of treatment, choosing the most suitable material for each patient and following the manufacturer's instructions for their cementing and adhesion.

SUMMARY:
A record of the type of onlay will be made with respect to its extension, tooth or teeth to be treated, the material of clothing and the substrate on which the adhesion and cementing method, as well as the type of antagonist. To complete it, a complete clinical oral examination will be performed with oral mirrors, examination probes, joint paper, disposable gloves, masks, paper napkins, plastic cups, dental equipment lighting lamp, cold spray , photogrammed camera, including an intraoral scan to have a 3D file of the patient's condition on the day of embedding placement.

Once treatment is complete, the patient should go to routine check-ups in which a full intraoral exploration and data collection intended to be carried out analyze the following variables (USPHS modificated): possible decemented and fractured, decay and marginal integrity, sensitivity or loss of vitality, as well as the degree of patient satisfaction (VAS).

DETAILED DESCRIPTION:
The same intervention will be carried out during the duration of the project, collecting the variables:

* baseline recall. (cementing day)
* 1 month.
* 6 months.
* annually.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Healthy adult patients (ASA I) susceptible to treatment with onlays in the posterior region treated at the University Dental Clinic (Master's Clinic in Dental Prosthetics of the Department of Stomatology of the Faculty of Medicine and dentistry)

Exclusion Criteria:

* Minor patients.
* Medically committed patients.
* Patients with active cavities.
* Patients with active periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Survival | Through study completion, an average of 5 years.
  Analyze the survival over time of this type of treatment

SECONDARY OUTCOMES:
Complications | Through study completion, an average of 5 years.
  Analyze complications over time of this type of treatment using modified UPSHS criteria

OTHER OUTCOMES:
Clinical behaviour | Through study completion, an average of 5 years.
  Analyze clinical behavior taking into account possible variables that may influence using modified UPSHS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Fernandez-Estevan, Doctor, Principal Investigator — University of Valencia
Locations (1):
- Lucia Fernandez-Estevan, Valencia, Spain